CLINICAL TRIAL: NCT06916013
Title: Transperineal Targeted Focal Laser Ablation of Localized Intermediate Risk Prostatic Adenocarcinoma (Pilot Study)
Brief Title: Focal Laser Ablation in Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: Laser in prostate cancer
Record Dates: First submitted 2025-02-14; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Laser
Keywords: Prostate cancer; Laser
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prostatic adenocarcinoma: Localized intermediate-risk prostatic adenocarcinoma
  Interventions: Procedure: Focal laser ablation

INTERVENTIONS:
Procedure: Focal laser ablation — Targeted focal laser ablation
Procedure: Focal laser ablation — Targeted focal laser ablation of localized intermediate-risk prostate cancer

SUMMARY:
To assess the effectiveness of MRI-US or PSMA PET/CT-U/S fusion-guided focal laser ablation (FLA) for the treatment of a localized, intermediate-risk prostate cancer in terms of short-term oncological & functional outcomes.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the second most common neoplasm diagnosed in men with an estimated 1.4 million diagnoses and 375,000 deaths worldwide in 2020.

For localized prostate cancer (PCa), active surveillance (AS) or whole gland treatment (ie, radical prostatectomy [RP] and radiotherapy) are considered standard treatment options. Unfortunately, treatment-related morbidity is high.

The ProtecT trial showed urinary incontinence rates of 3% and 20% and erectile dysfunction rates of 66% and 79% for radiotherapy and radical prostatectomy, respectively. Radiotherapy can also cause rectal problems with a small increased risk of radiotherapy-induced secondary malignancy.

Consequently, over the past few years, there has been a notable escalation in scholarly attention towards the implementation of focal therapeutic interventions for patients diagnosed with low- and intermediate-risk prostate cancer (PCa).

This tissue-preserving strategy has at its core the reduction of treatment-related toxicity by minimizing damage caused to the prostate and adjacent structures while attempting to retain the benefits of treating cancer.

The rationale of focal therapy (FT) is based on the theory that the largest lesion with the highest grade, the so-called "index lesion," determines the risk of metastases and thus the patient's prognosis.

FT involves ablating only the index lesion, thereby minimizing damage to collateral tissue such as neurovascular bundles, external urinary sphincter, bladder neck and rectum.

Over the past few years, different types of energy sources in FT have been studied. These consist of high-intensity focused ultrasound (HIFU), irreversible electroporation (IRE), cryotherapy, photodynamic therapy (PDT), focal laser ablation (FLA) or laser interstitial thermotherapy, radiofrequency ablation (RFA), and focal brachytherapy.

According to the European Association of Urology (EAU), low-risk and intermediate-risk patients may undergo local procedures using HIFU or cryotherapy within clinical trials or registries, with the aim of achieving long-term cancer control and reducing morbidity associated with surgery and radiation therapy.

Many groups have published limited data on outcomes following in-bore MRI-guided focal therapy, and many others are actively engaged or considering prospective comparative effectiveness research in this area.

The primary objective encompasses a thorough evaluation of the short-term oncological & functional outcomes of MRI-US or PSMA PET/CT-U/S fusion-guided focal laser ablation (FLA) for the treatment of a small, localized, intermediate-risk prostate cancer.

Concurrently, the secondary aim involves an assessment of the utility of multiparametric magnetic resonance imaging (mpMRI) as a diagnostic pre-treatment tool and during the post-treatment follow-up to examine the morphostructural alterations in the prostate gland resulting from FLA. Additionally, the investigatirs aim to assess its reproducibility in determining the response to FLA therapy, correlating these findings with biopsy results, with the ultimate objective of establishing its predictive diagnostic value in identifying residual or recurring tumors.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer visible on mpMRI or PSMA PET/CT and positive in the targeted biopsy.
* Gleason score 7 (ISUP grade 2/3)
* PSA 10-20 ng/mL
* Clinical stage T2b
* Refusing radical prostatectomy.

Exclusion Criteria:

* Prostate cancer invisible on mpMRI or PSMA PET/CT but positive in the systematic biopsies.
* Presence of >2 MRI-visible lesions and positive in the biopsies.
* Extracapsular extension
* Seminal vesicle invasion
* Presence of metastases detected by imaging
* Gleason Score > 7
* Stage > T2b
* PSA > 20 ng/mL
* Urinary tract infection (UTI)
* Severe lower urinary tract symptoms defined as an IPSS >20
* Severe coagulation disorders
* Inadequate compliance
* Contraindications to MRI
* Paramagnetic contrast agent allergy
* Acute and/or chronic renal failure

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Males with localized, intermediate risk prostatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of short-term oncological outcome | 12 months
  Follow-up with clinical evaluation performed by mpMRI. mpMRI is done for assessment of tissue changes as well as residual or recurrent disease after 10 days, then after 3 months, after 6 months then every 6 months thereafter.

SECONDARY OUTCOMES:
Evaluation of functional outcome. | 12 months
  IIEF-5 questionnaire is submitted at 3, 6, 12 months.

REFERENCES:
- [Result] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Result] Valerio M, Cerantola Y, Eggener SE, Lepor H, Polascik TJ, Villers A, Emberton M. New and Established Technology in Focal Ablation of the Prostate: A Systematic Review. Eur Urol. 2017 Jan;71(1):17-34. doi: 10.1016/j.eururo.2016.08.044. Epub 2016 Aug 29. PMID 27595377
- [Result] Ahmed HU. The index lesion and the origin of prostate cancer. N Engl J Med. 2009 Oct 22;361(17):1704-6. doi: 10.1056/NEJMcibr0905562. No abstract available. PMID 19846858
- [Result] Eggener S, Salomon G, Scardino PT, De la Rosette J, Polascik TJ, Brewster S. Focal therapy for prostate cancer: possibilities and limitations. Eur Urol. 2010 Jul;58(1):57-64. doi: 10.1016/j.eururo.2010.03.034. Epub 2010 Mar 26. PMID 20378241
- [Result] Lindner U, Trachtenberg J, Lawrentschuk N. Focal therapy in prostate cancer: modalities, findings and future considerations. Nat Rev Urol. 2010 Oct;7(10):562-71. doi: 10.1038/nrurol.2010.142. Epub 2010 Sep 14. PMID 20842187
- [Result] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Result] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338

DOCUMENTS (1):
  • Study Protocol (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT06916013/Prot_000.pdf